CLINICAL TRIAL: NCT02808208
Title: A Phase I, Open Label, Randomized Study of Autologous Adipose Derived Mesenchymal Stem Cells (AMSC) in Reducing Hemodialysis Arteriovenous Fistula Failure
Brief Title: Autologous Adipose Derived Mesenchymal Stem Cells (AMSC) in Reducing Hemodialysis Arteriovenous Fistula Failure
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sanjay Misra, M.D., M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-009053
Record Dates: First submitted 2016-06-02; First posted 2016-06-21 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease (ESRD); Vascular Access Complication
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single dose AMSC treatment in Radiocephalic (RCF)or brachiocepahlic (BCF) arteriovenous fistula (Experimental): Subjects who receive a radiocephalic (RCF)or brachiocepahlic (BCF) arteriovenous fistula through standard of care procedure for dialysis, will receive a single dose of Autologous Adipose Derived Mesenchymal Stem Cells (AMSC)
  Interventions: Biological: Single Application of Adipose Derived Mesenchymal Stem Cells (AMSC)
- No Treatment in Radiocephalic (RCF)or brachiocepahlic (BCF) arteriovenous fistula (No Intervention): Patients receive standard of care.
- Single dose AMSC treatment at first stage of brachiobasilic arteriovenous fistula (Experimental): Subjects who receive a brachiobasilic arteriovenous fistula (BBF) through standard of care procedure for dialysis, will receive a single dose of Autologous Adipose Derived Mesenchymal Stem Cells (AMSC) at time of first stage of BBF
  Interventions: Biological: Single Application of Adipose Derived Mesenchymal Stem Cells (AMSC)
- AMSC treatment at first and second stage of brachiobasilic arteriovenous fistula (Experimental): Subjects who receive a brachiobasilic arteriovenous fistula (BBF) through standard of care procedure for dialysis, will receive Autologous Adipose Derived Mesenchymal Stem Cells (AMSC) at first and second stage of BBF
  Interventions: Biological: Two Applications of Adipose Derived Mesenchymal Stem Cells (AMSC)
- Placebo treatment in brachiobasilic arteriovenous fistula (Placebo Comparator): Subjects will receive placebo at first and second stage of BBF
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Single Application of Adipose Derived Mesenchymal Stem Cells (AMSC) — A single topical application of mesenchymal stem cells derived from own fat biopsy to the surface of the outflow vein (right next to the fistula) over a five-minute period.
  Arms: Single dose AMSC treatment at first stage of brachiobasilic arteriovenous fistula; Single dose AMSC treatment in Radiocephalic (RCF)or brachiocepahlic (BCF) arteriovenous fistula
Drug: Placebo — 5-mL of Lactated Ringers solution topical application to the surface of the outflow vein (right next to the fistula) over a five-minute period.
  Arms: Placebo treatment in brachiobasilic arteriovenous fistula
Biological: Two Applications of Adipose Derived Mesenchymal Stem Cells (AMSC) — Two topical applications of mesenchymal stem cells derived from own fat biopsy to the surface of the outflow vein (right next to the fistula) over a five-minute period at stage one and two of fistula surgery
  Arms: AMSC treatment at first and second stage of brachiobasilic arteriovenous fistula

SUMMARY:
The aim of this phase 1 study is to determine the role of autologous adipose derived mesenchymal stem cells in the reduction of hemodialysis arteriovenous fistula failure when applied during the time of surgical creation.

ELIGIBILITY:
Inclusion Criteria

* Patient between 18 and 85 years old
* Patient currently on hemodialysis or pre-dialysis and planned creation of an upper extremity AV fistula with suitable anatomy
* Ability to communicate meaningfully with investigative staff, competence to give written informed consent, and ability to comply with entire study procedures
* Life expectancy of at least 24 months

Exclusion Criteria

* Malignancy or treatment for malignancy within the previous 6 months
* Immunodeficiency including AIDS / HIV or Active autoimmune disease
* Documented hypercoagulable state or history of 2 or more DVTs or other spontaneous intravascular thrombotic events
* Pregnancy or breast feeding
* Treatment with any investigational drug/ device within 60 days prior to study entry or Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of AMSCs and the AVF
* Employees of the sponsor or patients who are employees or relatives of the investigator
* History of failed organ transplant on immunosuppression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hemodialysis outflow vein diameter | Baseline to 12 months after AVF creation
  Diameter of outflow vein by ultrasound

SECONDARY OUTCOMES:
Hemodialysis AVF Blood flow | Baseline to 12 months after AVF creation
  blood flow by ultrasound or dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Misra, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piryani AK, Kilari S, Takahashi E, DeMartino RR, Mandrekar J, Dietz AB, Misra S. Rationale and Trial Design of MesEnchymal Stem Cell Trial in Preventing Venous Stenosis of Hemodialysis Vascular Access Arteriovenous Fistula (MEST AVF Trial). Kidney360. 2021 Sep 28;2(12):1945-1952. doi: 10.34067/KID.0005182021. eCollection 2021 Dec 30. PMID 35419530
- See also: Mayo Clinic Clinical Trials — http://ClinicalTrials.gov